CLINICAL TRIAL: NCT05483270
Title: Immediate Versus Postponed Freeze-all Embryo Transfer in Hyperresponders, a Multicenter Randomised Controlled Trial
Brief Title: Immediate Versus Postponed Freeze-all Embryo Transfer in Hyperresponders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: Women's Hospital School Of Medicine Zhejiang University (Other); The Affiliated Hospital Of Guizhou Medical University (Other); Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Li Rong, Professor, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Delay-ET-RCT
Record Dates: First submitted 2022-07-20; First posted 2022-08-02 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2023-05

CONDITIONS: IVF

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate FET group (Active Comparator): Freeze-all embryo transfer will be carried out in the menstrual cycle immediately following oocyte retrieval.
  Interventions: Biological: the timing of embryo transfer in freeze-all cycles
- Postponed FET group (Experimental): Freeze-all embryo transfer will be carried out during the second menstrual cycle to 6 months after oocyte retrieval.
  Interventions: Biological: the timing of embryo transfer in freeze-all cycles

INTERVENTIONS:
Biological: the timing of embryo transfer in freeze-all cycles — Immediate FET group Freeze-all embryo transfer will be carried out in the menstrual cycle immediately following oocyte retrieval.
  Postponed FET group Freeze-all embryo transfer will be carried out during the second menstrual cycle to 6 months after oocyte retrieval.

SUMMARY:
This is a multicenter, randomised controlled trial. The investigators plan to randomise 836 participants to the immediate FET or the postponed FET from the day of oocyte retrieval to the last day of that menstrual cycle in a 1:1 rate. Primary outcome will be the live birth rate after the embryo transfer.

DETAILED DESCRIPTION:
It is postulated that postponing embryo transfer for at least one menstrual cycle after a freeze-all cycle can minimise the possible residual negative effect caused by ovarian stimulation and can promote the resumption of a normal ovulatory cycle and the receptivity of endometrium. Nevertheless, emerging evidence suggests a higher live birth rate in the immediate freeze-all embryo transfer (FET) cycles compared to that in the delayed group. It is unclear the whether postponed FET is superior in hyperresponders. The investigators hypothesize the success rate in the postponed FET for at least one menstrual cycle after oocyte retrieval is higher than in the immediate FET in hyperresponders.

Objective: To evaluate whether the postponed FET for at least one menstrual cycle after oocyte retrieval is superior to the immediate FET in the first menstrual cycle after oocyte retrieval in hyperresponders in terms of live birth rates.

Design: a multicenter, randomised controlled trial Patients: The investigators plan to randomise participants to the immediate FET and the postponed FET from the day of oocyte retrieval to the last day of that menstrual cycle.

Primary outcome: live birth rate after the embryo transfer. Patients who get pregnant will be followed up until 6 weeks after delivery.

Sample size: The investigators plan to enroll 836 participants in a 1:1 rate.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 20 to 42 years old;
* Written informed consent;
* Women scheduled for freeze-all embryo transfer;
* Women with the number of oocyte collected higher than 15.

Exclusion Criteria:

* Women with a history of at lease three failed transfer cycles;
* Women with an endometrial thickness less than 7 mm on the triggering day;
* Severe uterine malformations.

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 845 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-11-24 (Actual)

PRIMARY OUTCOMES:
Live birth after the first embryo transfer | At least 22 months gestation after the first embryo transfer cycle
  Live birth is defined as the delivery of at least one baby after 22 weeks of gestation that exhibits any sign of life.

SECONDARY OUTCOMES:
Clinical pregnancy | around 7 weeks' gestation after the first embryo transfer cycle
  defined as at least one gestational sac on ultrasound at around 7 weeks' gestation with the detection of heart-beat activity
Ongoing pregnancy | 12 weeks' gestation or beyond after the first embryo transfer cycle
  defined as pregnancy with detectable heart rate at 12 weeks' gestation or beyond
Biochemical pregnancy | about 12 days after embryo transfer
  defined as a positive pregnancy test
Ectopic pregnancy | about 6 weeks after embryo transfer
  defined as embryo implanted at any site other than the endometrial lining of the uterus cavity
Miscarriage | 6-22 weeks of gestation
  defined as spontaneous loss of a clinical pregnancy before 22 completed weeks of gestational age, in which the embryo(s) or fetus(es) is/are nonviable or is/are absorbed or expelled from the uterus.
Cumulative live birth | 6 month after the first embryo transfer
  the cumulative rate of live born children conceived within six months of the first FET cycle.
Pre-eclampsia | after 20 weeks of gestation
  defined as the development of gestational hypertension with proteinuria (≥300 mg/24-hour urine collection or 30 mg/dL in single urine sample) of new onset after 20 weeks of gestation
Gestational hypertension | after 20 weeks of gestation
  defined as the development of blood pressure greater than 140/90 mmHg after pregnancy without proteinuria or other signs of preeclampsia
Gestational diabetes mellitus | after 24 weeks of gestation
  defined as carbohydrate intolerance of variable severity with onset or first recognition during pregnancy as determined from the diagnosis in the obstetrical medical record
Premature rupture of membrane (PROM) rate | the day of delivery
  defined as rupture of the amniotic membranes before the onset of labor including PROM at term and preterm PROM
Preterm delivery | less than 37 and more than 21 weeks' gestational age
  defined as delivery of a fetus at less than 37 weeks' gestational age
Placenta previa | the day of delivery
  defined as a placenta that is implanted over or very close to the internal cervical orifice
Postpartum hemorrhage | the day of delivery
  defined as the loss of 500 ml of blood or more after completion of the third stage of labor
Birth weight | the day of delivery
  Birth weight
Stillbirth | the day of delivery
  defined as the absence of signs of life at or after birth
Mode of delivery | the day of delivery
  Vaginal birth or Caesarean Section

CONTACTS AND LOCATIONS:
Overall Officials: Kai-Lun Hu, M.D, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking university third hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Results of the study will be submitted to scientific conferences in reproductive medicine and a peer-reviewed journal.
Supporting Information: Study Protocol, SAP
Time Frame: The day of publishing the main results. Around 3 years from now
Access Criteria: Please contact the hukailun@bjmu and roseli001@sina.com